CLINICAL TRIAL: NCT06132048
Title: A Usability Validation of the MuCopilot Mobile Application, a Digital Tool for the Unsupervised Objective Assessment of Cystic Fibrosis
Acronym: MuControl-Sum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ad scientiam (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADS-MuControl-Summative-2023
Record Dates: First submitted 2023-10-31; First posted 2023-11-15 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MuCopilot - Summative evaluation (Experimental): Performance of digital tests and questionnaire from MuCopilot, during the visit.
  Interventions: Device: MuCopilot mobile application

INTERVENTIONS:
Device: MuCopilot mobile application — MuCopilot is a software as medical device with three digital tests, to measure patient's with CF, lung function, global exercise capacity and a questionnaire to address CF symptoms and impacts on some aspects of patient's life

SUMMARY:
The study aims to assess the usability and safety of use of MuCopilot, a smartphone application that measures objective data on lung function, global exercise capacity and patient reported outcomes of patients with Cystic Fibrosis (CF). These data are collected during unsupervised digital tests performed in the patient's home environment between consultations.

The primary objective is to validate the usability and safety of use, in order to assure that the patients use the medical device as intended without any unacceptable error of use and without unacceptable risk.

The study will include 17 CF patients and will be conducted in France. They will participate in 1 inclusion visit and 1 visit in-clinic (1h30).

Patients will be able to download the free MuCopilot mobile application. During the visit, patients will complete 3 digital tests in order to monitor CF functions (cough, dyspnea & walking) and 1 symptom questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Aged ⩾ 18 years old
* Patients diagnosed with cystic fibrosis
* Enrolled in or benefiting of a Social Security program
* Having read the information sheet and signed the informed consent form
* Owning a personal smartphone which version is above 14 for IOS and 8 for Android included with a good internet connexion
* Able to read French and understand pictograms on a smartphone app

Exclusion Criteria:

* History of lung transplantation
* Pregnant women and women who are breastfeeding
* Any medical condition that could interfere with the proper conduct and results of the study (clinician's judgement)
* Illiterate in French
* Inability to use a smartphone or MuCopilot application
* Person under legal protection (including guardianship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Validation of usability (1) | 2 hours
  Use error : Any deviation from the instructions for use that does not result in a response from the medical device other than what the manufacturer intended. Validated if there is no unacceptable use error.
Validation of usability (2) | 2 hours
  Task completion rate: percentage of use scenarios completed without observation of an unacceptable error. The unacceptable nature of an error is determined according to the risk analysis process covered by ISO 14971:2019. Validated if the success rate on each task must reach 78% at minimum.
Validation of no safety critical of use | 2 hours
  Safety critical error: a user error that causes a safety incident, where safety is defined as the appearance of a hazardous situation and the related harms linked to an unacceptable risk, as stated in the application version of Risk Analysis. Validated if there is no safety critical error has been identified during the evaluation.
Validation of ease of use | 2 hours
  The MuCopilot solution will be considered as easy to use, if the perceived ease of use" mean score reaches 7.8/10

CONTACTS AND LOCATIONS:
Locations (1):
- CRCM Mixte - Hôpital Charles Nicolle, Rouen, France

IPD SHARING:
Plan to Share IPD: No